CLINICAL TRIAL: NCT02508402
Title: Effect Of Intra-muscular Administration of Dexamethasone on the Duration of Induction of Labour in Primigravida Post-term Pregnancy.
Brief Title: Effect Of Intra-muscular Administration of Dexamethasone in Induction of Labour
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed El-Sharkawy, Lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KasrELAiniH
Record Dates: First submitted 2015-07-14; First posted 2015-07-24 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-09

CONDITIONS: Medical Induction of Labor Affecting Fetus
MeSH Terms: interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexamethasone group (Active Comparator): The participant of Dexamethasone Group will receive a prefilled syringe with two milliliters (8 mg) of Dexamethasone intramuscular After six hours of the initial dose, the labour induction will start via Oxytocin .III. The interval between the initiation of induction and the beginning of the active phase of labour is recorded (a cervical dilatation of 4 cm plus 3 forceful contractions over a 10-minute span each last from 40-60 Sec).
  Interventions: Drug: Dexamethasone
- Placebo group (Placebo Comparator): and the participants of placebo Group will not receive Dexamethasone or any other cervical ripening agent.II.two milliliters of normal saline given.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — The participant of Dexamethasone Group will receive a prefilled syringe with two milliliters (8 mg) of Dexamethasone intramuscular, and the participants of Group II will not receive Dexamethasone or any other cervical ripening agent.
  All the participants in both groups will randomly be assigned by computer list.
  II. After six hours of the initial dose, the labour induction will start via Oxytocin using
  Other Names: epidrone
  Arms: dexamethasone group
Drug: Placebo — two milliliters of normal saline given to placebo group .
  Other Names: Normal saline
  Arms: Placebo group

SUMMARY:
ABSTRACT:

Objective: To evaluate the efficacy of dexamethasone on labor duration and to establish whether dexamethasone plays a role in shorting the duration interval between initiation of labor induction and beginning of the active phase in primigravida full-term pregnancy.

Methods: case control study included 86 primigravidae with full term pregnancy classified into two groups: The participant of Group I will receive a prefilled syringe with two milliliters (8 mg) of Dexamethasone intramuscular, and the participants of Group II will not receive Dexamethasone or any other cervical ripening agent.

Key Words: Dexamethasone;post-term pregnancy;induction of labor.

DETAILED DESCRIPTION:
METHODS:

This retrospective clinical trial was conducted at the Department of Obstetrics and Gynecology, Faculty of Medicine, Cairo University, during the period from August 2014 to May 2015. The study protocol was approved by the Scientific Research Committee, and informed consent was obtained from all participants.

Each participant will randomly be assigned by computer list into Group I (Dexamethasone group(n=43)and group II(control group(N=43).

No cervical ripening agent will be used for induction of labour in the trial.

Methodology in details:

I. The participant of Dexamethasone Group will receive a prefilled syringe with two milliliters (8 mg) of Dexamethasone intramuscular, and the participants of placebo Group will not receive Dexamethasone or any other cervical ripening agent.

All the participants in both groups will randomly be assigned by computer list. (Haijavandi et., al 2013)

II. After six hours of the initial dose, the labour induction will start via Oxytocin using the following protocol:

1. Initial dose of oxytocin.................................. 1 to 2 milliliter international unit/min.
2. Increase interval......................................................30 minutes.
3. Dosage increment....................................................1 to 2 milliliter international unit/min.
4. Usual dose for good labour.........................8 to12 milliliter international unit/min.
5. Maximum dose…………………...................30 milliliter international unit/min. (Anne Biringer et., al 2013).

III. The interval between the initiation of induction and the beginning of the active phase of labour is recorded (a cervical dilatation of 4 cm plus 3 forceful contractions over a 10-minute span each last from 40-60 Sec).

IV. Partographic representation for progression of active phase labour:

1. Frequency and duration of uterine contraction.
2. Cervical dilatation will record every two hours by per vaginal examination.
3. Station and position of fetal head was noted at the same time.

V. After delivery:-

1. The duration of the first stage of labor will be recorded. (Partographic representation will do for each participant).
2. The duration of the second stage of labor will be recorded.
3. The duration of the placental separation will be recorded.
4. The neonatal outcome will be recorded by APGAR score.
5. Any postpartum maternal adverse effect was noted (e.g. vital sign abnormality, any maternal postpartum hemorrhage).

Primary outcome:

the duration between induction and beginning of active phase.

Secondary outcome:

-Duration of first stage.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Primigravida.
* Post-term gestation i.e. 41 weeks or more.
* Sure, reliable dates.
* Favorable cervix with Bishop score of 7 or greater.
* Longitudinal lie.
* Cephalic presentation (Vertex).

Exclusion Criteria:

* Abnormal presentation.
* Multigravida.
* Multiple pregnancies.
* Active phase of labour.
* Cephalo-pelvic disproportion.
* History of any medical disorder.
* History of previous myomectomy operation.
* Known contraindication or hypersensitivity to Dexamethasone.
* Current fetal distress.
* Current maternal or fetal disorder e.g. Diabetes mellitus; Pregnancy induced hypertension, and fetal growth retardation.
* Over distended abdomen e.g. fetal macrosomia or polyhydramnios suggested by ultrasound or estimated fetal weight by expert hand.
* Significant vaginal bleeding.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
the duration between induction and beginning of active phase. | 6 months

SECONDARY OUTCOMES:
Duration of first stage. | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Abdel Aziz El Sharkawy, Cairo, Egypt